CLINICAL TRIAL: NCT05394753
Title: The Efficacy of Group-based Unified Protocol (UP) Programme for Improving Sleep and Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EA210411
Record Dates: First submitted 2022-02-14; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Quality of Life; Insomnia; Depression, Anxiety
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unified Protocol (Experimental): 8-session group-based intervention
  Interventions: Behavioral: Unified Protocol for mood disorders
- Wait-list control (No Intervention): Participants in the wait-list control group will receive the same program, two months after their counterparts in the experimental group completed the intervention.

INTERVENTIONS:
Behavioral: Unified Protocol for mood disorders — The group-based UP is structured and manualized and consists of 9 1.5 hours weekly sessions (90-min, 18 participants in each group). The group-based UP is a course consisting of components of psycho-education about mood disorders, cognitive and behavioural skills, and relapse prevention and is adapted for the non-clinical population in the current study. The UP will be led and delivered by trained therapists.
  Arms: Unified Protocol

SUMMARY:
Common mental disorders can be disabling and lead to a large burden of disease. Unified Protocol for Transdiagnostic Treatment of Emotional Disorders was developed to address emotional disorders with evidence-based emotional-focused cognitive-behavioural techniques and is efficacious in reducing anxiety symptoms and depressive symptoms in adults. Previous research has demonstrated comparable effect of UP on reducing anxiety symptoms compared with the single-disorder protocol (SDP) for anxiety. Group-based UP was also implemented and tested. Given the fact that working populations are at a high risk of poor mental health, especially in light of the COVID pandemic with new unprecedented work situations and increased uncertainties, the present study aims to investigate the efficacy of Unified protocol on sleep and mental health in high-risk population.

ELIGIBILITY:
Inclusion Criteria:

* Working in local schools or education institutions
* aged 18 or above
* no severe or unstable mental health conditions at recruitment
* no extensive prior training/practice with mindfulness

Exclusion Criteria:

* psychotic disorders, bipolar disorder, severe alcohol disorder and substance abuse, acute and high suicidal risk
* currently receiving taking other psychosocial interventions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change in Positive affect | week 1, week 5, week 9, 12 weeks after completion of intervention
  Positive and Negative Affect Schedule (PANAS), 4 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Negative affect | week 1, week 5, week 9, 12 weeks after completion of intervention
  Positive and Negative Affect Schedule (PANAS), 4 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change of insomnia symptoms | week 1, week 5, week 9, 12 weeks after completion of intervention
  Insomnia symptoms are measured by Insomnia Severity Index (ISI). ISI is a 5-item self-rated scale. Possible scores range from 0 to 20, with higher scores indicating higher insomnia severity.

SECONDARY OUTCOMES:
Change of Sleep Diary Measure - Time in Bed (TIB) | week 1, week 9, 12 weeks after completion of intervention
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: time in bed (TIB) in hours
Change of Sleep Diary Measure - Total Sleep Time (TST) | week 1, week 9, 12 weeks after completion of intervention
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: total sleep time (TST) in hours
Change of Sleep Diary Measure - Sleep Onset Latency (SOL) | week 1, week 9, 12 weeks after completion of intervention
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep onset latency (SOL) in mins
Change of Sleep Diary Measure - Wake After Sleep Onset (WASO) | week 1, week 9, 12 weeks after completion of intervention
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: wake after sleep onset (WASO) in mins
Change of Sleep Diary Measure - Sleep Efficiency (SE) | week 1, week 9, 12 weeks after completion of intervention
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %
Change in Objective Sleep Measures - Time in Bed (TIB) | week 1, week 9, 12 weeks after completion of intervention
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: time in bed (TIB) in hours
Change in Objective Sleep Measures - Total Sleep Time (TST) | week 1, week 9, 12 weeks after completion of intervention
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: total sleep time (TST) in hours
Change of objective sleep measure (sleep onset latency, SOL) | week 1, week 9, 12 weeks after completion of intervention
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep onset latency (SOL) in mins
Change in Objective Sleep Measures - Wake After Sleep Onset (WASO) | week 1, week 9, 12 weeks after completion of intervention
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: wake after sleep onset (WASO) in mins
Change in Objective Sleep Measures - Sleep Efficiency (SE) | week 1, week 9, 12 weeks after completion of intervention
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %
Change in General Health | week 1, week 5, week 9, 12 weeks after completion of intervention
  General Health Questionnaire (GHQ), 12 items, 4-point Likert scale ranging from 1 (never) to 5 (always)
Change in Stress | week 1, week 5, week 9, 12 weeks after completion of intervention
  Perceived Stress Scale (PSS), 10 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Compassion | week 1, week 9, 12 weeks after completion of intervention
  Compassion scale, 6 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Self-compassion | week 1, week 9, 12 weeks after completion of intervention
  Self-compassion scale, 6 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Common humanity | week 1, week 9, 12weeks after completion of intervention
  Common Humanity scale, 10 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Mindfulness | week 1, week 9, 12 weeks after completion of intervention
  Cognitive and Affective Mindfulness Scale-Revised (CAMS-R), 12 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Decentering | week 1, week 9, 12 weeks after completion of intervention
  Non Reactivity Subscale of Chinese Five Facet Mindfulness Questionnaire (FFMQ-C), 4 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Emotion Regulation | week 1, week 5, week 9,12 weeks after completion of intervention
  Reappraisal subscale of Emotion Regulation Questionnaire (ERQ), 10 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change of clinically depressive symptoms | week 1, week 5, week 9, 12 weeks after completion of intervention
  Patient Health Questionnaire-9 (PHQ-9) consists of 9 self-report items designed to assess clinically significant depression. Higher scores indicate high level of depression.
Change of clinically anxiety symptoms | week 1, week 5, week 9, 12 weeks after completion of intervention
  General Anxiety Disorder-7 (GAD-7) consists of 7 self-report items designed to assess general anxiety symptoms. Higher scores indicate high level of anxiety.
Change of subjective mental well-being | week 1, week 5, week 9, 12 weeks after completion of intervention
  The World Health Organisation- Five Well-Being Index (WHO-5) consists of 5 self-report items designed to measure subjective well-being. Higher scores indicate better well-being.
Change of pre-sleep arousal | week 1, week 9, 12 weeks after completion of intervention
  Pre-Sleep Arousal Scale is a 16-item self-rated scale measuring pre-sleep arousal. There are two subscales on the cognitive and somatic manifestations of arousal, with eight items in each subscale (possibly scored from 8 to 40). In both cases, a higher score indicates higher pre-sleep arousal.
Change of sleep reactivity | week 1, week 9, 12 weeks after completion of intervention
  Ford Insomnia Response to Stress Test (FIRST) consists of 9 items designed to measure sleep reactivity. Possible scores range from 9 to 36. A higher score indicates higher sleep activity.
Change of quality of life | week 1, week 5, week 9, 12weeks after completion of intervention
  WHOQOL-BREF, 26 items, 5-point Likert scale ranging from 1 (never/very bad/strongly disagree) to 5 (always/very good/strongly agree)
TMSS-repair | week 1, week 9, 12 weeks after completion of intervention
  Trait Meta-Mood Scale repair subscale, 6 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
RRS | week 1, week 5, week 9, 12 weeks after completion of intervention
  Ruminative responsive scale, 22 items, 4-point Likert scale ranging from 1 (almost never) to 4 (almost always)

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Research Clinic and Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong